CLINICAL TRIAL: NCT01634659
Title: Clinical Evaluation of Two Daily Disposable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M-12-033
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Myopia
Keywords: contact lenses; myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delefilcon A, then narafilcon B (Other): Delefilcon A contact lenses (DAILIES TOTAL1®) worn first, followed by narafilcon B contact lenses (1-DAY ACUVUE® TruEye®). Each product was worn bilaterally (ie, in both eyes) in a daily wear, daily disposable mode for 8 days.
  Interventions: Device: Delefilcon A contact lenses (DAILIES TOTAL1®); Device: Narafilcon B contact lenses (1-DAY ACUVUE® TruEye®)
- Narafilcon B, then delefilcon A (Other): Narafilcon B contact lenses (1-DAY ACUVUE® TruEye®) worn first, followed by delefilcon A contact lenses (DAILIES TOTAL1®). Each product was worn bilaterally (ie, in both eyes) in a daily wear, daily disposable mode for 8 days.
  Interventions: Device: Delefilcon A contact lenses (DAILIES TOTAL1®); Device: Narafilcon B contact lenses (1-DAY ACUVUE® TruEye®)

INTERVENTIONS:
Device: Delefilcon A contact lenses (DAILIES TOTAL1®) — Commercially marketed silicone hydrogel, single-vision contact lenses for daily wear, daily disposable use
Device: Narafilcon B contact lenses (1-DAY ACUVUE® TruEye®) — Commercially marketed, silicone hydrogel single-vision contact lenses for daily wear, daily disposable use

SUMMARY:
The purpose of this study was to compare the subjective performance of DAILIES TOTAL1® daily disposable contact lenses to that of 1-DAY ACUVUE® TruEye® daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Sign written Informed Consent Document and HIPAA form.
* Be current weekly/monthly replacement contact lens wearer.
* Be willing to not sleep in contact lenses during the study period.
* Require vision correction in both eyes, with a contact lens prescription in protocol-specified power range.
* Have best corrected visual acuity of at least 20/25 in each eye.
* Be willing to wear study lenses for at least 8 hours/day and at least 5 days/week.
* Use re-wetting drops less than once per day and be willing to discontinue use of rewetting drops while wearing the study contact lenses.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Be a neophyte or current wearer of daily disposable lenses.
* Require monovision correction or use multifocal contact lenses.
* Have any systemic or ocular disease or disorder, complicating factor, or structural abnormality that would negatively affect the conduct or outcome of the study.
* Have a history of ocular surgery/trauma within the last 6 months.
* Use topical ocular or systemic antibiotics within 7 days of enrollment.
* Use topical ocular or systemic corticosteroids within 14 days of enrollment, continuing throughout the study.
* Have participated in any other ophthalmic drug or device clinical trial within 30 days of enrollment.
* Have habitually worn contact lenses on an extended wear basis (sleeping in habitual contact lenses for at least 2 nights per week) in the last 3 months prior to enrollment.
* Use re-wetting drops once or more per day.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, MBA, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 18 study centers located in the US.
Pre-assignment Details: Of the 330 participants enrolled, 17 were exited from the study prior to randomization and dispense of product.This reporting group includes all randomized and dispensed participants (313).
Period: Period 1 - First 8 Days of Wear
Arm/Group | Delefilcon A, Then Narafilcon B | Narafilcon B, Then Delefilcon A
Started | 155 | 158
Completed | 155 | 158
Not Completed | 0 | 0
Period: Period 2 - Second 8 Days of Wear
Arm/Group | Delefilcon A, Then Narafilcon B | Narafilcon B, Then Delefilcon A
Started | 155 | 158
Completed | 152 | 158
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized and dispensed participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Delefilcon A, Then Narafilcon B | Narafilcon B, Then Delefilcon A | Total
Number analyzed (Participants) | 155 | 158 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (10.0) | 32.1 (8.8) | 32.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 120 | 237
  Male | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort was interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 8 days of wear. Overall comfort was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent. Both eyes contributed to the mean.
Time Frame: Day 8
Population: Per-Protocol: All participants completing the study and satisfying all of the inclusion/exclusion criteria, minus protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Delefilcon A: Delefilcon A contact lenses (DAILIES TOTAL1®) worn bilaterally in a daily wear, daily disposable mode for 8 days in either Period 1 or Period 2
- Narafilcon B: Narafilcon B contact lenses (1-DAY ACUVUE® TruEye®) worn bilaterally in a daily wear, daily disposable mode for 8 days in either Period 1 or Period 2
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 301 | 301
Units on a scale | 8.5 (1.7) | 8.6 (1.5)

2. Secondary Outcome: Overall Quality of Vision
Description: Overall quality of vision was interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 8 days of wear. Overall quality of vision was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent. Both eyes contributed to the mean.
Time Frame: Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 301 | 301
Units on a scale | 8.6 (1.6) | 8.5 (1.6)

3. Secondary Outcome: End of Day Comfort
Description: End of day comfort was interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 8 days of wear. End of day comfort was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent. Both eyes contributed to the mean.
Time Frame: Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Narafilcon B
Number analyzed (Participants) | 301 | 301
Units on a scale | 7.7 (2.2) | 7.9 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (3 months).
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the study medical device. This reporting group includes all randomized and dispensed participants.
Arm/Group | Delefilcon A | Narafilcon B
Serious Adverse Events (participants affected / at risk) | 0/313 | 0/313
Other Adverse Events (participants affected / at risk) | 0/313 | 0/313

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.